CLINICAL TRIAL: NCT07055204
Title: Multicenter Study Evaluating the Efficacy of a Cognitive Remediation Method Using Rhythmic, Vocal and Corporal Musical Learning for Schizophrenia Patients
Brief Title: Cognitive Remediation Method Using Rhythmic, Vocal and Corporal Musical Learning for Schizophrenia
Acronym: ARCoS-2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC31/24/0332
Record Dates: First submitted 2025-06-12; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Schizophrenia Disorders
Keywords: cognitive remediation; music; rythmic; vocal; corporal; musical learning
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Intervention Model Description: national, multicenter, randomized, open label, comparative study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Diapason & Metronome" musical learning arm (Experimental): The "Diapason & Metronome" musical learning method was developed specifically by the authors of the study. Participants will make music with the two instruments we all have in common: the voice and the body.
  Interventions: Other: "Diapason & Metronome" musical learning
- standard of care arm (No Intervention): Patients randomly assigned in the control group will receive standard regular outpatient psychiatric care with at least one therapeutic or social activity (except musical or rhythmic activities).
  The "standard of care" is defined by regular psychiatric follow-up by a doctor specialised in psychiatry, and the use of antipsychotic medication. Care may be provided by a private psychiatrist, a Centre Médico-Psychologique (CMP) or a psychiatric day hospital. The frequency of treatment can vary from weekly to monthly, depending on the patient's state of stability. In addition, patients must be enrolled in at least one social or therapeutic activity during the week (therapeutic workshop in a day hospital or CATTP (Centre Accueil Thérapeutique à Temps Partiel), workshop in a GEM (Groupe d'Entraide Mutuelle), voluntary activity, club sport, or professional activity).

INTERVENTIONS:
Other: "Diapason & Metronome" musical learning — Participants will make music with the two instruments we all have in common: the voice and the body. The method is three-dimensional built on: rhythm, simple sound and harmony. The music sessions will take place in the same place and on the same day of the week, at a fixed time to establish a regularity that is suitable to this population. The courses will be taught in a cultural location, both to give meaning to the approach on a contextual level and to allow patients to be in the city and not in the hospital. A training of the music teachers will be planned before the beginning of the study. This training combined with regular debriefings during the music sessions, should ensure that the teachers' practices are consistent across the different groups.
  Arms: "Diapason & Metronome" musical learning arm

SUMMARY:
Schizophrenia, affecting 1% of the population, is a persistent disorder characterized by varied symptoms. Antipsychotic medications effectively address positive symptoms (delusions, hallucinations) and relapse but have limited impact on negative symptoms (e.g., blunted affect, anhedonia) and cognitive impairment. These dimensions significantly influence social functioning and quality of life. Combining non-pharmacological approaches like Cognitive Remediation (CR) and psychosocial rehabilitation alongside antipsychotic drugs is recommended to enhance overall functioning and quality of life. Current CR programs show moderate effectiveness due to patient commitment issues. However, completed programs demonstrate higher efficacy. Real-life applicability of these programs lacks sufficient data. We propose musical learning for cognitive remediation due to its established cognitive benefits in the general population, targeting executive functions, working memory, attention, and inhibition. These functions are specifically impaired in schizophrenia and thus are relevant for remediation. Though unexplored in schizophrenia, music learning seems promising due to its motivational and pleasurable aspects for long-term commitment and its transferability through embodied and situated dimensions. A pilot study (ARCoS-1) on CR by musical learning demonstrated feasibility and preliminary positive results on cognitive and negative symptoms. This project aims to assess this method's effectiveness on a larger scale. Our hypothesis posits that musical learning offers an efficient and well-received medium for CR in patients with schizophrenia.

DETAILED DESCRIPTION:
This study will be a national, multicenter, randomized, open label, comparative study evaluating the impact of 6-month collective embodied musical learning program on attentional deficits, in comparison with a control group receiving standard care.

Patients will be randomized in each center in 2 groups: one group will participate in weekly musical learning sessions, the other one will beneficit of standard care.

The study will be conducted in 2 phases:

* Phase 1 (six months of collective rhythmic, vocal and corporal musical training): 6 groups of 10 patients will participate in 6-month collective musical training provided by a professional music teacher. Sessions will start no later than 3 months after the inclusion, at the rate of one session per week for a period of 6 months (24 sessions in all, as part of a pedagogical project). Each session lasts one hour.
* Phase 2: a post-remediation follow-up period of 3 months (after the musical training sessions have stopped) to evaluate the potential lasting effect of group musical training on cognitive disorders and negative symptoms in patients.

For each patient, the duration of the protocol is 9 months, with assessment visits scheduled at regular 3-month intervals (Inclusion, M3, M6 and M9) for a total of 4 visits. Before the inclusions begin, 6 music teachers will be trained in the musical learning method developed for this project (one teacher in each participating town : Bayonne, Lyon, Marseille, Paris, Toulouse).

ELIGIBILITY:
Inclusion Criteria:

* Patient with a diagnosis of schizophrenia or schizoaffective disorder (DSM-5 TR criteria)
* Clinically stable (no full-time hospitalization related to schizophrenia for 3 months)
* Regular psychiatric follow-up
* Enrolled in at least 1 therapeutic or social out-of-home activity
* No change in the antipsychotic treatment for 3 months (medication and/or dosage)
* Have given free, informed and written consent to participate in the study.
* Patient affiliated or beneficiary of a social security scheme

Exclusion Criteria:

* Patient with moderate to severe intellectual disability (clinical criteria)
* Engaged in a Social rythmic or musical activity
* Presenting an addictive comorbidity (excluding tobacco addiction and behavioural addictions)
* Presenting a neurological pathology with cognitive impact
* Involved in a neurocognitive remediation program

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01-04 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
attention capacity | Baseline = Day 0 ; Month 6
  The primary endpoint will be to compare treated and control groups on the change from baseline to M6 (evaluation at the end of the remediation phase) of the D2-R scale score.
  D2-R scale (Brickenkamp, R. et al, 2015) is a paper-and-pencil test that provides a fine-tuned measure of selective and sustained attention.
  The test requires the subject to identify and cross out target characters (d with 2 dashes) from a large number of distractor characters. It therefore requires concentrated and sustained visual attention, and mobilises inhibitory control. There are three indicators of the strategy employed and the evolution of concentration:
  * CC - concentration capacity or concentration performance
  * CCT - work rhythm or processing speed
  * E% - processing precision --> the higher the score for each category, the better the attention capacity is

SECONDARY OUTCOMES:
Attentional deficits at 3 months after the start of the remediation (M3) and at 3 months post-remediation (M9) | Baseline = Day 0 ; Month 6 and Month 9 (evaluation at 3 month of the remediation phase)
  Change from baseline to M3 and M9 (evaluation at 3 month of the remediation phase) of the D2-R scale score
  D2-R scale (Brickenkamp, R. et al, 2015) is a paper-and-pencil test that provides a fine-tuned measure of selective and sustained attention.
  The test requires the subject to identify and cross out target characters (d with 2 dashes) from a large number of distractor characters. It therefore requires concentrated and sustained visual attention, and mobilises inhibitory control. There are three indicators of the strategy employed and the evolution of concentration:
  * CC - concentration capacity or concentration performance
  * CCT - work rhythm or processing speed
  * E% - processing precision --> the higher the score for each category, the better the attention capacity is
Attentional phasic alert at 3 months after the start of remediation (M3), at the end of the remediation phase (M6) and at 3 months post-remediation (M9). | Baseline = Day 0 ; Month 6 and Month 9
  Change in attention abilities evaluated by the results obtained in the phasic alert test of the TAP, from baseline to M3, M6 and M9.
  TAP = Test of Attentional Performance is a computer-based battery for assessing attention. The phasic alert test : refers to a state of general arousal that allows for quick and appropriate responses to stimuli. It is an indispensable condition for effective behavior and constitutes, from this point of view, a basis for all attentional performances. Reaction times (RT) are examined under two conditions. The first concerns the evaluation of simple RT: a cross appears in the center of the screen after randomly varying inter-stimulus intervals, and the subject must react as quickly as possible by pressing a response key. In this condition, intrinsic alertness is measured. In the second condition, RTs are measured as responses to the same cross but this time preceded by a (auditory) stimulus.
  --> The lowest the RT, the better is the attention ability

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - CH de la Côte Basque, Bayonne
  - CH Le Vinatier, Bron
  - Assistance Publique Hôpitaux de Marseille, Marseille
  - Association route nouvelle, Toulouse
  - Centre de Santé MGEN, Toulouse
  - CH Gérard Marchant, Toulouse

IPD SHARING:
Plan to Share IPD: No